CLINICAL TRIAL: NCT07063264
Title: Effects of High-definition Transcranial Direct Current Stimulation During Slow-wave Sleep on Associative Memory
Brief Title: Effects of HD-tDCS During Slow-wave Sleep on Associative Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WANG KAI (Other)
Responsible Party: Sponsor-Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HD-tDCS-healthy adults
Record Dates: First submitted 2025-06-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Transcranial Direct Current Stimulation; Healthy Adults
Keywords: Associative Memory; High-Definition Transcranial Direct Current Stimulation; Slow Wave Sleep; DLPFC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sleep with active stimulation (Sleep-A) (Active Comparator): Participants will receive active anode HD-tDCS during slow-wave sleep (SWS) of non-rapid eye movement sleep (NREM) at afternoon nap. An anode stimulation electrode will be placed in F3 (10/20 system) which intended to target the left DLPFC, and four cathodes will be placed at FCz, AFz, F7, and C5 (10/20 system)
  Interventions: Device: high-definition transcranial direct current stimulation (HD-tDCS)
- sleep with sham stimulation (Sleep-S) (Placebo Comparator): Participants will receive afternoon nap with sham stimulation. A 30-s rising current until 2 mA is reached, with a 30-s decline immediately at the beginning and end of the stimulation section
  Interventions: Device: sham high-definition transcranial direct current stimulation (HD-tDCS)
- wake with active stimulation (Wake-A) (Sham Comparator): Participants will receive active anode HD-tDCS during wakefulness. They will receive HD-tDCS stimulation for 25 minutes while awake, then spent free time in the sleep monitoring room, remaining awake throughout the napping period
  Interventions: Device: high-definition transcranial direct current stimulation (HD-tDCS)

INTERVENTIONS:
Device: high-definition transcranial direct current stimulation (HD-tDCS) — HD-tDCS is described as a non-invasive form of brain stimulation that uses a low-intensity, direct current applied directly to the head through scalp electrodes
  Arms: sleep with active stimulation (Sleep-A); wake with active stimulation (Wake-A)
Device: sham high-definition transcranial direct current stimulation (HD-tDCS) — Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Arms: sleep with sham stimulation (Sleep-S)

SUMMARY:
To evaluate the effects of afternoon naps and high-definition transcranial direct current stimulation (HD-tDCS) over the left dorsolateral prefrontal cortex (DLPFC) in associative memory (AM)

DETAILED DESCRIPTION:
Healthy adults will be randomized into three groups: a sleep with active stimulation (Sleep-A) group will receive active anode HD-tDCS during slow-wave sleep (SWS) of non-rapid eye movement sleep (NREM) at afternoon nap, a sleep with sham stimulation (Sleep-S) group will receive afternoon nap with sham stimulation, and wake with active stimulation (Wake-A) group will receive active anode HD-tDCS during wakefulness. An anode stimulation electrode will be placed in F3 (10/20 system) which intend to target the left DLPFC, and four cathodes will be placed at FCz, AFz, F7, and C5 (10/20 system). The face-word AM task and other multidimensional neuropsychological tasks will be performed before and after afternoon napping.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-30 years
* healthy adults

Exclusion Criteria:

* with pacemakers, skull cavities or cracks；
* intolerance of high-definition transcranial direct current stimulation (HD-tDCS) adverse reactions；
* left-handed；
* diagnosed with severe mental disorders, or involved in other experiments.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
face-word assciative memory task score | 1 hour after the end of the afternoon nap
  In the face-cued word association test, participants viewed 20 grayscale photographs of faces on a computer screen, each shown for 3 seconds. Each photograph was paired with a distinct word, which participants read aloud when shown. Participants were instructed to memorize the word linked to each face. One minute later, participants viewed the same 20 faces in a new random order. They were then asked to recall the associated words. Each face was scored as correct or incorrect, and the total number of correct responses formed the AM score.

SECONDARY OUTCOMES:
Auditory Verbal Learning Test (AVLT) score | 2 hours after the end of afternoon nap
  There are two parts to the test process: learning phase and delayed recall phase. During the learning phase, subjects were asked to listen to a list of words and recall them. During the delayed recall phase, subjects were asked to recall the list of previously learned words again after a period of time. Scoring usually includes recording the number of correct memories the subject has during the learning phase and delayed recall phase, as well as the types of possible errors (such as forgetting, confusion, etc.). Depending on the subject's performance, learning and memory abilities can be assessed. The normal ranges of immediate memory, delayed memory and recognition memory were 10, 8 and 10 respectively. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China